CLINICAL TRIAL: NCT05344599
Title: Estimating the Frequency and Neuro-Hormonal Characteristics of Acute Hepatic Porphyria in Postural Tachycardia Syndrome
Brief Title: Evaluating the Prevalence of Acute Hepatic Porphyria in Postural Tachycardia Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Associate Professor, Vanderbilt University Medical Center
Other Study IDs: 210724
Record Dates: First submitted 2022-04-08; First posted 2022-04-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Postural Orthostatic Tachycardia Syndrome; Acute Hepatic Porphyria
Keywords: POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Coproporphyria, Hereditary | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood, Serum Urine, Saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Autonomic Function Testing — Autonomic function test (orthostatic blood pressure and heart rate response to tilt, heart rate response to deep breathing, the Valsalva ratio, and beat-to-beat blood pressure measurements during phases II and IV of the Valsalva maneuver, tilt, and deep breathing). These combined tests provide a measurement of adrenergic, cardiovagal responses.
Diagnostic Test: Genetic Testing — Genetic testing: for Acute hepatic porphyria panel - with intent to use Saliva kit
Diagnostic Test: Urine Testing — Urine PBG, ALA and porphyrins in a spot urine sample with results normalized to urine creatinine
Diagnostic Test: Blood laboratory Testing — To determine the following laboratory analyses:
  CBC, CMP, Iron studies (Ferritin and iron studies)

SUMMARY:
Postural Tachycardia Syndrome (POTS) is the most common autonomic disorder and is estimated to affect 3,000,000 individuals in the United States, with 80-85% of patients being women. The condition is characterized by a rapid increase in heart rate (HR) that occurs on standing, and chronic symptoms of cerebral hypoperfusion leading to lightheadedness, dizziness, and blurred vision.

The acute hepatic porphyrias(AHP)are among the diseases that present with autonomic cardiovascular(tachycardia)and neurovisceral symptoms (abdominal pain) among others; they present with acute exacerbations Given that there is available treatment for AHP that change the natural progression of the disease, study focuses to investigate the occurrence of AHP in POTS and determine the clinical and neuro-hormonal characteristic of the POTS subgroup that will likely benefit from AHP screening.

This study has one visit that involves, answering some questionnaires, coming to the lab for blood work, genetic testing, and some autonomic function tests. About 50 people will take part in this study.

DETAILED DESCRIPTION:
Postural Tachycardia Syndrome (POTS) affects ~3 million young women in the United States.(1)These patients have a low quality of life because of chronic presyncopal symptoms, and orthostatic tachycardia that occur while standing. POTS can be the initial presentation of an underlying illness. A substantial group of patients with POTS reported that their symptoms started after an acute illness, surgical intervention, substantial weight loss or after ingesting certain medications. These are the same triggers for acute AHP attacks.

Furthermore, the demographic characteristics of AHP overlaps with that of POTS. AHP also affects primarily young women, in their reproductive age. POTS can have a diverse presentation, some patients present with axonal autonomic neuropathy, and severe gastrointestinal symptoms which are co-morbid conditions also present in chronic AHP.

It is within this context that investigators propose to assess the occurrence of AHP in the general POTS population, identify its clinical presentation and neuro-hormonal characteristics.

Rationale and Endpoints:

1. To evaluate occurrence of AHPs in POTS patients with autonomic and neurovisceral symptoms referred to a National Referral Center for the treatment of Autonomic Disorder.
2. To determine the autonomic and neuro-hormonal characteristics of AHP-POTS patients compared with POTS patients

Enrollment:

This is a cross-sectional study conducted at the Vanderbilt Autonomic Dysfunction Clinic (ADC). Investigators plan to enroll patients with suspicions of POTS who are referred to the ADC for evaluation and diagnosis.

Study visit:

Single study visit.

Participants will be asked to complete an autonomic symptoms assessment questionnaire (COMPASS 31), and quality of life EQ-5D.

The following laboratory analyses will be performed:

Blood: CBC, CMP, Iron studies (Ferritin and iron studies) Urine PBG, ALA and porphyrins in a spot urine sample with results normalized to urine creatinine.

Genetic testing (Acute hepatic porphyria panel) .

Autonomic function test.

Supine and Standing plasma norepinephrine will be obtained for evaluation of neuro-hormonal changes during orthostasis.

Statistical Analyses

This is a pilot study that will estimate the occurrence of AHPs in POTS patients referred to a National Referral Center for the Treatment of Autonomic Disorders. There is no data available on the prevalence of AHPs in POTS. The prevalence of AHP is one in 6,000 in whites. [ref. Hepatol commun 2019 feb 3(2): 193-206] Given that there are overlapping of symptoms between AHP and POTS, expected that AHP would be overrepresented in POTS patients. The plan is to enroll 50 POTS patients in this pilot study.

Data Analysis Plan:

Standard graphing and screening techniques will be used, to detect outliers and to ensure data accuracy. Continuous endpoints will be assessed for normality. If normality is violated, data transformation will be applied or non-parametric analysis methods will be considered. Investigators will provide summary statistics for both continuous and categorical variables by subject groups (POTS and AHP-POTS). All hypotheses will be tested, at the level of α=0.05. SPSS (version 23.0, SPSS, Chicago, IL) will be used and the open-source statistical package R (R Core Team, 2019 for analyses.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 - 65 years
2. Individuals having an established diagnosis of POTS defined as the presence of presyncopal symptoms for more than 6 months and orthostatic tachycardia (>30 bpm increase in HR within 10 min after assuming upright position)
3. The present of one of the following criteria:

3.1 Family history of acute hepatic porphyria 3.2 Unexplained recurrent (more than one), prolonged (>24 hours) episode of severe, diffuse (poorly localized) abdominal pain AND at least TWO of the following:

* Red to brownish urine.
* Blistering skin lesions on sun-exposed areas.
* Peripheral nervous system manifestations occurring around the time of abdominal pain (i.e., motor neuropathy (paresis), sensory neuropathy (numbness, tingling, limb pain).
* Central nervous system manifestations occurring around the time of abdominal pain (i.e. confusion, anxiety, seizures, hallucinations).
* Autonomic nervous system manifestations occurring around the time of abdominal pain (i.e. hyponatremia(Na<lower limit of normal)), tachycardia, hypertension, nausea and vomiting, constipation).

Exclusion Criteria

1. Pregnant or breastfeeding women
2. type 2 diabetes mellitus
3. History of alcohol or drug abuse
4. Inability to provide informed consent or comply with protocol

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes, gender self-identity
Study Population: Postural Tachycardia Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
AHP Case ascertainment in POTS patients | During the intervention
  Evaluating the Prevalence of Acute Hepatic Porphyria in Postural Tachycardia Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, M.D, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robertson D. The epidemic of orthostatic tachycardia and orthostatic intolerance. Am J Med Sci. 1999 Feb;317(2):75-7. doi: 10.1097/00000441-199902000-00001. No abstract available. PMID 10037110
- [Result] Garland EM, Raj SR, Black BK, Harris PA, Robertson D. The hemodynamic and neurohumoral phenotype of postural tachycardia syndrome. Neurology. 2007 Aug 21;69(8):790-8. doi: 10.1212/01.wnl.0000267663.05398.40. PMID 17709712
- [Result] Schondorf R, Low PA. Idiopathic postural orthostatic tachycardia syndrome: an attenuated form of acute pandysautonomia? Neurology. 1993 Jan;43(1):132-7. doi: 10.1212/wnl.43.1_part_1.132. PMID 8423877
- [Result] Raj SR. The Postural Tachycardia Syndrome (POTS): pathophysiology, diagnosis & management. Indian Pacing Electrophysiol J. 2006 Apr 1;6(2):84-99. PMID 16943900
- [Result] Loavenbruck A, Iturrino J, Singer W, Sletten DM, Low PA, Zinsmeister AR, Bharucha AE. Disturbances of gastrointestinal transit and autonomic functions in postural orthostatic tachycardia syndrome. Neurogastroenterol Motil. 2015 Jan;27(1):92-8. doi: 10.1111/nmo.12480. Epub 2014 Dec 6. PMID 25483980